CLINICAL TRIAL: NCT05389384
Title: The Effect of a Passive Shoulder Exoskeleton and Muscle Fatigue on Occupational Work Performance
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Romain Meeusen, Principle Investigator, Vrije Universiteit Brussel
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Prevention
Other Study IDs: 2021_E4W_SH_PER
Record Dates: First submitted 2021-04-26; First posted 2022-05-25 (Actual); Last update posted 2022-05-25 (Actual); Status verified 2022-05

CONDITIONS: Fatigue; Muscle Strain; Physical Stress
Keywords: peripheral fatigue; overhead work; task performance; ergonomics; effort
MeSH Terms: conditions — Fatigue; Sprains and Strains

STUDY DESIGN:
Intervention Model Description: counterbalanced randomized cross-over study
Who Masked: Participant
Masking Description: The support of the exoskeleton is concealed. The support will be 'no support' or 'support'.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Peripheral fatigue - No support (Experimental): peripheral fatigue induced and overhead work performed without exoskeleton support
  Interventions: Behavioral: Fatigue protocol; Device: No exoskeleton support
- Peripheral fatigue - Exoskeleton support (Experimental): peripheral fatigue induced and overhead work performed with exoskeleton support
  Interventions: Device: Passive shoulder exoskeleton; Behavioral: Fatigue protocol
- No fatigue - No support (Experimental): peripheral fatigue induced and overhead work performed without exoskeleton support
  Interventions: Device: No exoskeleton support; Behavioral: No peripheral fatiguing protocol
- No fatigue - Exoskeleton support (Experimental): peripheral fatigue induced and overhead work performed with exoskeleton support
  Interventions: Device: Passive shoulder exoskeleton; Behavioral: No peripheral fatiguing protocol

INTERVENTIONS:
Device: Passive shoulder exoskeleton — Participants complete overhead working task with support of exo
  Arms: No fatigue - Exoskeleton support; Peripheral fatigue - Exoskeleton support
Behavioral: Fatigue protocol — Participants complete a fatiguing protocol
  Arms: Peripheral fatigue - Exoskeleton support; Peripheral fatigue - No support
Device: No exoskeleton support — Exoskeleton is worn, but no support provided
  Arms: No fatigue - No support; Peripheral fatigue - No support
Behavioral: No peripheral fatiguing protocol — Participants complete no fatiguing protocol
  Arms: No fatigue - Exoskeleton support; No fatigue - No support

SUMMARY:
In this investigation, participants perform simulated occupational work during which the task performance will be logged. This research investigates the effect of peripheral fatigue and a passive shoulder exoskeleton on the task performance.

ELIGIBILITY:
Inclusion Criteria:

* healthy (based on ParQ questionnaire)
* right handed

Exclusion Criteria:

* current musculoskeletal disorder
* history of recurrent musculoskeletal discorder

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2021-08-20 (Actual); Primary Completion 2022-07-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Work accuracy | During 2 minutes overhead work
  The number of errors is tracked
Work pace | During 2 minutes overhead work
  Time to completion is tracked

SECONDARY OUTCOMES:
Surface electromyography | During 2 minutes overhead work
  Cometa (Mini Wave) sensors with Ambu (BlueSensor) electrodes will be used to collect electromyographic data conform the SENIAM guidelines. The muscles that will be monitored are: deltoideus anterior, deltoideus medialis, deltoideus posterior, pectoralis major, latissimus dorsi, brachioradialis, biceps brachii, triceps brachii, trapezius descendens, infraspinatus, supraspinatus, flexor carpi radialis, serratus anterior on the right side of the body. The locations of the sensors will be prepared by shaving, abrasion with sandpaper and cleaning with alcohol. To allow relative expression of muscle activity, maximal voluntary contractions (MVC) of each muscle that is being monitored will be collected. The average of the maximal activity out of the best two out of three contractions will serve as the MVC value. The outcomes will be the activities of the muscles (as a percentage of the MVC) monitored during the tests.
Kinematic smoothness of movement | During 2 minutes overhead work
  Inetrial Measurement Units will be used to track how smoothly the overhead work is completed. Smoothness is determined by the Spectral Arc method.
Workload | After 2 minutes of overhead work
  NASA TLX questionnaire for workload

OTHER OUTCOMES:
Force output | before and after 4 minute during fatigue inducing protocol
  measure output force during elevation of the arms in a 45° flexed shoulder angle

CONTACTS AND LOCATIONS:
Overall Officials: Romain Meeusen, PhD, Principal Investigator — Vrije Universiteit Brussel
Locations (1):
- Lichamelijk Opvoeding en Kinesitherapie, Brussels, Belgium

IPD SHARING:
Plan to Share IPD: No
Data will be published in scientific journal. No IPD will be published.